CLINICAL TRIAL: NCT05552170
Title: Evaluation of Short-term Outcomes of Ambulatory Loop Ileostomy Reversal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Colorectal Cancer Center, Department of General Surgery, West China Hospital
Other Study IDs: DS-2017
Record Dates: First submitted 2022-09-19; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Surgery; Fast Recovery Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- day case group: Patients who underwent loop ileostomy with age ≤ 65 and ASA II or III were enrolled and underwent ALIR after rigorous evaluation.
  Interventions: Other: day-case surgery

INTERVENTIONS:
Other: day-case surgery — Patients who underwent loop ileostomy with age ≤ 65 and ASA II or III were enrolled and underwent ALIR after rigorous evaluation.

SUMMARY:
Based on enhanced recovery after surgery (ERAS), ambulatory loop ileostomy reversal (ALIR) has been reported in developed countries. However, there is still no research proposing how to carry out ALIR in developing countries. This study was performed to determine the feasibility of ALIR in China based on the community hospital joined enhanced recovery after surgery (CHJ-ERAS) program.

DETAILED DESCRIPTION:
CHJ-ERAS program for ALIR was launched. Patients who underwent loop ileostomy with age ≤ 65 and ASA II or III were enrolled and underwent ALIR after rigorous evaluation. Strict follow-ups were conducted after ALIR. The primary outcome was the results of short-term follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ileostoma and preparing for LIR
2. Patients age between 18-65;
3. ASA grade II;
4. Patients willing to underwent day-case LIR

Exclusion Criteria:

* 1) Patients who underwent single-lumen ileostomy, transverse colostomy or Hartmann; 2) Complex previous laparotomies or required exploratory laparotomy; 3) Age over 65; 4) ASA grade over III (assessed by anesthetists); 5) Presence of moderate or severe preoperative anemia (hemoglobin <90g/L); 6) Therapeutic anticoagulation or anti-platelet medications used within 1 week before surgery; 7) Patient refusal; 8) Severe co-morbidities or other conditions evaluated by surgeons or anesthetists not inappropriate to be included in the program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All potential patients preparing for LIR were asked to undergo multiple evaluations at our outpatient department by gastrointestinal surgeons and anesthetists together. They were admitted to our ambulatory surgery center and included in the CHJ-ERAS program for ALIR if none of the exclusion criteria was met.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Results of short-term follow-up | Within 1 month after surgery
  The occurrence of postoperative complications
Readmissions | Within 1 month after surgery
  Readmission within 1 month after surgery
Reoperation | Within 1 month after surgery
  Reoperation within 1 month after surgery

SECONDARY OUTCOMES:
Hospital stays | 1 day
  Hospital stays

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided